CLINICAL TRIAL: NCT00372931
Title: A Phase II Study of AL-37807 to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-06-15
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

INTERVENTIONS:
Drug: AL-37807

SUMMARY:
The purpose of this study is to determine whether AL-37807 is safe and effective in treating patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex and any race with open-angle glaucoma or ocular hypertension; logMAR visual acuity not worse than 0.60; additionally clinically relevant ophthalmic or systemic conditions may be excluded

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-05; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean IOP change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Study Director — Study Director
Locations (1):
- San Antonio Site, San Antonio, Texas, United States